CLINICAL TRIAL: NCT02280031
Title: Effect of Low Dose Aspirin on Birthweight in Twins: The GAP Trial
Acronym: GAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014-1817
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2016-04

CONDITIONS: Small for Gestational Age; Infant, Very Low Birth Weight; Fetal Growth Retardation; Preeclampsia; Premature Birth
Keywords: Twin Pregnancy; Pregnancy Complications
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia; Premature Birth; Pregnancy Complications | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Active Comparator): Acetylsalicylic Acid 80mg administered daily at bedtime
  Interventions: Drug: Acetylsalicylic Acid
- Control (Placebo Comparator): Identical placebo administered daily at bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic Acid — Capsule containing Acetylsalicylic Acid 80mg pill with lactose
  Other Names: Aspirin; ASA; Asaphen
  Arms: Experimental
Drug: Placebo — Capsule containing placebo pill with lactose
  Other Names: Control
  Arms: Control

SUMMARY:
Low-dose aspirin started in the first-trimester has been associated with a decrease of preeclampsia, fetal growth restriction and preterm birth in high-risk pregnancies. Multiple pregnancies are considered a risk factor for all those adverse outcomes. The main objective of the current trial is to evaluate whether a dose of 80 mg of aspirin is associated with an improvement of birthweight compared to placebo in twin pregnancies.

DETAILED DESCRIPTION:
Twin pregnancies represent approximately 3% of births and are associated with increased risks of complications such as preeclampsia, fetal growth restriction and preterm birth. All of these complications are commonly associated impaired placental function and low birth weight.

Most prophylactic measures tested over the years have failed to prevent these adverse outcomes in twin pregnancies. Since administration of low-dose of aspirin can improve placental function and all these adverse outcomes in high-risk pregnancies, mainly in women with prior adverse outcomes, we suggest that similar benefits could be seen in twins. We are expecting that the administration of low-dose of aspirin starting in the first-trimester in twin pregnancies could lead to an improvement of placental function, a reduction or these adverse perinatal outcomes and therefore to an improvement of birthweight.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 8 0/7 and 13 6/7 weeks
* Twin pregnancy confirmed by ultrasound

Exclusion Criteria:

* One or two negative heart beat
* Previous hypertensive disorder of pregnancy
* Pre-existing hypertension or diastolic blood pressure >90 mmHg at randomization
* Pre-existing nephropathy
* Pre-existing diabetes (type 1 or 2)
* Anaphylactic allergy to lactose
* Known coagulopathy (antithrombin III deficiency, factor V Leiden, antiphospholipid syndrome, the prothrombin mutation, deficiency of protein S or protein C)
* Use of heparin or other anticoagulants.
* Contre-indications to aspirin
* Discordance of crown-rump length greater than 20%.
* Fetal anomalies (cystic hygroma, nuchal translucency > 95th percentile, anencephaly, omphalocele, etc.)
* Previous or current gastric ulcer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Birth weight | At delivery

SECONDARY OUTCOMES:
Low birth weight | At delivery
  (birthweight below 2,500 grams)
Very low birth weight | At birth
  (birthweight below 1,500 grams)
Fetal growth restriction | 16-18 and 22-24 weeks
  (birthweight below the 10th or 3rd percentile for gestational age)
Preterm birth | At delivery
  (delivery before 37 weeks)
Very preterm birth | At delivery
  (delivery before 34 weeks)
Preeclampsia | At delivery
  (according to American College of Obstetricians and Gynecologists 2014 guidelines definition)
Early-onset preeclampsia | At delivery
  (onset of preeclampsia before 34 weeks)
UtA_PI | 22-24 weeks
  Mean uterine artery pulsatility index
Aspirin resistance | 16-18 and 22-24 weeks
  (PFA-100 below 150)
Cervical length | 22-24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD,MSc,FRCSC, Principal Investigator — CHU de Québec
Locations (2):
- Canada (2):
  - Hôpital St-François d'Assise-CHUQ, Québec
  - Centre Hospitalier Universitaire de Québec (CHU de Québec)/Pavillon CHUL, Québec